CLINICAL TRIAL: NCT05236972
Title: Study of Sintilimab vs Standard Therapy in Participants With Mismatch Repair Deficient (dMMR) or Microsatellite Instability-High (MSI-H) Stage III Colorectal Cancer
Brief Title: PACE: PD-1 Antibody For dMMR/MSI-H Stage III Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); West China Hospital (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2021-361-01
Record Dates: First submitted 2022-01-19; First posted 2022-02-11 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Carcinoma
Keywords: dMMR/MSI-H
MeSH Terms: conditions — Colorectal Neoplasms | interventions — sintilimab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab (Experimental): Sintilimab 200mg iv drip Q3W for 8 courses
  Interventions: Drug: Sintilimab
- XELOX (Experimental): Patients receive chemotherapy comprising oxaliplatin 130mg/m² ivdrip over 2 hours on day 1,capecitabine 2000 mg/m² on days 1-14, treatment repeats every 21 days for 4 or 8 courses
  Interventions: Drug: Oxaliplatin; Drug: capecitabine

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg iv drip Q3W
  Arms: Sintilimab
Drug: Oxaliplatin — 130 mg/m² iv drip over 2 hours on day 1, repeated every 21 days.
  Arms: XELOX
Drug: capecitabine — 1000 mg/m² po twice daily on days 1- 14 repeated every 21 days
  Arms: XELOX

SUMMARY:
In this open-label phase III study, patients with local advanced colon cancer (TanyN+ ,M0, dMMR/MSI-H, at least 10cm from the anus verge)will be scheduled to Group A: receive anti-PD-1 antibody alone (8 cycles, 200mg iv drip Q3W) and Group B (4 or 8 cycles of XELOX: oxaliplatin 130mg/m2 day 1, capecitabine 2000mg/m2 days 1-14, repeated every 21 days). The primary endpoint was 3 Disease-free survival; analyses were done based on all patients with post-randomization data.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years
2. ECOG PS 0/1
3. Histologically proven, stage III (i.e., any T, N1 or N2, M0) adenocarcinoma of the colon (as defined by the presence of the inferior pole of the tumour above the peritoneal reflection - that is, at least 10 cm from the anal margin).
4. Fully surgically resected tumour with clear resection margins (i.e., >1 mm)
5. Locally confirmed defective mismatch repair (dMMR) tumour (as defined by the lack of staining on either the pre-operative biopsy samples or resection specimens of at least one of the following proteins: MLH1 (mutL homolog 1), MSH2 (mutS homologue 2), MSH6 (mutS homolog 6), PMS2
6. Absence of metastases as shown by post-operative CT scan
7. Absence of major post-operative complications or other clinical conditions that, in the opinion of the investigator, would contraindicate adjuvant chemotherapy

Exclusion Criteria:

1. Rectal tumours (as defined by the presence of the inferior pole of the tumour below the peritoneal reflection - that is, <15 cm from the anal margin).
2. Inability to start adjuvant chemotherapy within 12 weeks after surgery
3. Administration of neoadjuvant systemic chemotherapy or radiotherapy before surgical resection of colon cancer
4. Prior organ transplantation, including allogeneic stem-cell transplantation
5. Significant acute or chronic infections including, among others:

   known history of testing positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) positive test for HBV (Hepatitis B) surface antigen or anti-HCV (Hepatitis C) antibody and confirmatory HCV RNA test
6. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:
7. Subjects with diabetes type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible
8. Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤10 mg/day of prednisone or equivalent
9. Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable
10. Known severe hypersensitivity reactions to monoclonal antibodies (Grade ≥3 NCI-CTCAE v4.0), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
11. Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v4.0; however, alopecia and sensory neuropathy Grade ≤2 is acceptable unless oxaliplatin administration is planned as part of the adjuvant treatment
12. Pregnancy or lactation
13. Known alcohol or drug abuse
14. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication
15. Known history of colitis, pneumonitis and pulmonary fibrosis (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the 16.Investigator, might impair the subject's tolerance of trial treatment.

Any psychiatric condition that would prohibit the understanding or rendering of informed consent 17.Other invasive malignancy within 2 years except for non-invasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Free survival [ Time Frame: 3 years ] | Up to 5 years
  Disease-free survival (DFS) at 3 years. DFS is measured from the date of randomisation to the date of first relapse (radiological or clinical) or death from any cause.

SECONDARY OUTCOMES:
Overall Survival [ Time Frame: 5 years ] | Up to 5 years
  Overall survival (OS) at 5 years. OS is measured from the date of randomisation to date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No